CLINICAL TRIAL: NCT03341494
Title: A Randomized Phase II Study of Gefitinib Alone Versus Gefitinib Plus Thalidomide for Advanced Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor Activating Mutations
Brief Title: EGFR Mutation Positive NSCLC Patients With Gefitinib and Thalidomide
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG002
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: NSCLC Stage IV; Chemotherapy Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefitinib 250mg qd thalidomide 200mg qn (Experimental)
  Interventions: Drug: Thalidomide
- Gefitinib 250mg qd (Active Comparator)
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Gefitinib 250mg Thalidomide 200 MG

SUMMARY:
EGFR-TKIs are the standard first-line treatment option for EGFR-mutant NSCLC. After a randomized phase II trial, JO25567 was presented at 2014 ASCO, the synergistic effect of progression-free survival(PFS) could be expected when EGFR TKI, Gefitinib is combined with Antiangiogenesis agent thalidomide, Therefore Chinese data of treating EGFR mutation positive NSCLC patients with Gefitinib and thalidomide is significantly necessary for developing new standard treatment in first-line therapy in Chinese EGFR mutant NSCLC patients.

In this study, The investigators will investigate the efficacy and safety of Gefitinib and thalidomide combination compare to Gefitinib alone in Chinese EGFR-mutant NSCLC patients.

DETAILED DESCRIPTION:
EGFR-TKIs are the standard first-line treatment option for EGFR-mutant NSCLC. After a randomized phase II trial, JO25567 was presented at 2014 ASCO, the synergistic effect of progression-free survival(PFS) could be expected when EGFR TKI, Gefitinib is combined with Antiangiogenesis agent thalidomide, . Even Chinese and Japanese are classified as Asian based on location, the figure of Chinese is more tended to Western people due to the dietary life in recent years. However the incidence rate of EGFR mutation positive patients in Chinese is much higher than Western countries.

Therefore Chinese data of treating EGFR mutation positive NSCLC patients with Gefitinib and thalidomide is significantly necessary for developing new standard treatment in first-line therapy in Chinese EGFR mutant NSCLC patients.

In this study, The investigators will investigate the efficacy and safety of Gefitinib and thalidomide combination compare to Gefitinib alone in Chinese EGFR-mutant NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage IIIB & IV non-small cell lung cancer other than squamous cell carcinoma

  * Patients with one or more measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
  * Locally diagnosed sensitive EGFR mutation positive (Exon 19 deletion or L858R)
  * ECOG performance 0~1
  * Age ≥ 19 years and - No previous treatment

Adequate organ function by following:

* ANC ≥1,500/uL, hemoglobin ≥9.0g/dL, platelet ≥100,000/uL
* Serum bilirubin < 1 x UNL, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, If Liver metastasis, Serum bilirubin < 3 x UNL, AST (SGOT) and ALT (SGPT) < 5 x UNL
* Serum Cr ≤ 1 x UNL
* Patients who have had undergone radiotherapy are acceptable if patients meet all of the following criteria:

  * No history of irradiation to pulmonary tumor lesions.
  * In case of palliative irradiation to bone lesions in lung: at least 12 weeks must have passed at the date of registration since the last irradiation of the sites.
  * In case of irradiation to non-pulmonary sites: at least two weeks must have passed at the date of inclusion since the last irradiation of the sites
* At the time of registration, at least the following period has passed since last date of the prior therapy or procedure:

  * Surgery(including exploratory/ examination thoracotomy): 4 weeks
  * Pleural cavity drainage: 1 weeks
  * Pleurodesis without anti-neoplastic agents (inclusive of BRM such as Picibanil): 2 week
  * Biopsy accompanied by incision (including thoracoscopic biopsy): 2 week
  * Procedure for trauma (exclusive of patients with unhealed wound): 2 weeks
  * Transfusion of blood, preparation of hematopoietic factor: 2 week
  * Puncture and aspiration cytology: 1 week
  * Other investigational product: 4 weeks
* Written informed consent form

Exclusion Criteria:

* • Previous history of malignancy within 3 years from study entry except treated non-melanomatous skin cancer, uterine cervical cancer in situ, or thyroid cancer

  * Prior chemotherapy or systemic anti-cancer therapy for metastatic disease but postoperative adjuvant or neoadjuvant therapy of 6 months or more previously is allowed
  * Patients who received previous treatment for lung cancer with drugs
  * Symptomatic or uncontrolled central nervous system (CNS) metastases
  * Patients with increased risk of bleeding, clinically significant cardiovascular diseases, a history of thrombosis or thromboembolism in the 6 months prior to treatment, gastrointestinal problems, and neurologic problems
  * Any significant ophthalmologic abnormality
  * Pre-existing parenchymal lung disease such as pulmonary fibrosis
  * Known allergic history of Erlotinib or Bevacizumab
  * Interstitial lung disease or fibrosis on chest radiogram
  * Active infection, uncontrolled systemic disease (cardiopulmonary insufficiency, fatal arrhythmias, hepatitis)
  * Pregnant or nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to at least 36 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | through study completion, and average of 2 years
  Overall Response Rate
OS | From date of randomization until the date of death or date of last visit/contact, whichever came first, assessed to at least 36 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Gen lin, Principal Investigator — Fujian Cancer Hospital
Locations (2):
- China (2):
  - Fujian Cancer Hospital Radiation Oncology Department, Fuzhou, Fujian
  - Fujian cancer hospital, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: yes
Access Criteria: yes